CLINICAL TRIAL: NCT04965155
Title: Isatuximab and Autologous Hematopoietic Stem Cell Transplantation for Relapsed Multiple Myeloma Patients (Isabel Study)
Brief Title: A Trial for Relapsed Multiple Myeloma Patients (Isatuximab-dexamethasone)
Acronym: ISABEL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EMN Trial Office S.r.l. Impresa Sociale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISABEL
Record Dates: First submitted 2021-07-02; First posted 2021-07-16 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Isatuximab-dexamethasone pre and post transplant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isatuximab-Dexamethasone (Experimental): Isatuximab-Dexamethasone pre and post transplant in relapsed multiple myeloma patients.
  Interventions: Drug: Isatuximab-dexamethasone

INTERVENTIONS:
Drug: Isatuximab-dexamethasone — Isatuximab 10 mg/kg IV: 1,8,15 and 22 at cycle 1; days 1 and 15 at cycles 2-3 Dexamethasone 40 mg OS: 1,8,15 and 22 at cycle 1; days 1 and 15 at cycles 2-3

SUMMARY:
This is an open label phase II study designed to assess the efficacy and safety of the combination isatuximab-dexamethasone pre and post transplant in relapsed MM patients. Before enrolment, patients have already received a reinduction therapy, as per local protocols, in order to achieve an optimal cytoreduction. Since carfilzomib-based regimens (eg. carfilzomib-lenalidomide-dexamethasone or carfilzomib-dexamethasone) are the current standard in Italy, for uniformity the use of one of these combinations is recommended. However, any cytoreductive treatment, excluding anti-CD38 antibodies containing regimens, as per local practice, is acceptable. During this period, if necessary, it will be possible to mobilize and collect peripheral blood stem cells. After the pre-enrollment cytoreduction period (reinduction therapy), patients have achieved at least a PR according to IMWG Response criteria.

After study enrolment, patients will receive 3 courses of isatuximab in combination with dexamethasone; after cycle 3 patients will receive ASCT, that will be conditioned with melphalan and will be followed by reinfusion of cryopreserved autologous stem cells. At 2 months after ASCT, patients will start maintenance, consisting in the administration of isatuximab in combination with dexamethasone for 12 cycles. Starting from cycle 13 onwards, only isatuximab will be administered until progression or intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given voluntary written informed consent
2. Patient is willing and able to comply with the study visits and procedures required per protocol
3. Subject must have at least 18 and = 70 years of age
4. Patient has a life-expectancy = 3 months
5. Subject has received an ASCT in the first line of therapy with a progression/relapse after at least 24 months
6. Subject must have received any cytoreductive treatment, excluding anti-CD38 antibodies containing regimens, as per local practice for the first relapse, according to local guidelines. Carfilzomib-based combinations are recommended (eg. carfilzomib-lenalidomidedexamethasone or carfilzomib-dexamethasone). After the salvage duration phase (reinduction therapy), subject has achieved at least a PR according to IMWG Response criteria.
7. Subject must have documented relapsed MM as per IMWG criteria, and achieved at least a partial remission with treatments as per local guidelines
8. Subject must have at least 2.0 x 106 CD34+/Kg cryopreserved autologous stem cells
9. Subject must have an ECOG Performance Status score of 0, 1
10. Subject must have the following laboratory values:

    * Platelet count =50 x 109/L (=30 x 109 /L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to drug administration)
    * Absolute neutrophil count (ANC) = 1 x 109/L without the use of growth factors
    * Corrected serum calcium =14 mg/dL (3.5 mmol/L)
    * Alanine transaminase (ALT): = 3 x the ULN
    * Total bilirubin: = 2 x the ULN
    * Calculated or measured creatinine clearance: = 30 mL/minute
11. Female subjects are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * they are not females of childbearing potential (FCBP), OR
    * they are FCBP who have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting study medication and before each cycle of study treatment and must either commit to continue abstinence from heterosexual intercourse or apply a highly effective method of birth control during the intervention period and for at least 5 months after the last dose of study treatment. Of note: contraception duration should take also into consideration any backbone therapy
12. Male subjects must agree to use contraception on this protocol during the intervention period and for at least 5 months after the last dose of study treatment and refrain from donating sperm during this period

Exclusion Criteria:

1. Previous therapy with daratumumab, isatuximab or any other anti-CD38 monoclonal antibody
2. MM localization to the central nervous system
3. Subjects who have received any investigational drug within 14 days or 5 half-lives of the investigational drug from eligibility confirmation, whichever is longer
4. Subjects who have received an allogeneic stem cell transplant
5. Subject with a history of malignancy (other than multiple myeloma) within 3 years before the date of eligibility confirmation (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, in agreement with the medical monitor, is considered cured with minimal risk of recurrence within 3 years)
6. Subject is known to be seropositive for human immunodeficiency virus (HIV) or with an active hepatitis A, B and C infection, defined as a positive test for hepatitis B surface antigen [HBsAg] and a positivity for HAV-RNA, HBV-DNA or HCV-RNA
7. Subject with any concurrent, clinically significant, uncontrolled medical condition or disease (eg, active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study
8. Subject with active tuberculosis and severe infections requiring treatment with an antibiotic parenteral administration
9. Subject with hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study therapy that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents
10. Subject with pulmonary deficit, defined as FEV1 <65% and/or DLCO <65%
11. Subject with clinically significant cardiac disease, including:

    * LVEF <50%
    * Myocardial infarction within 6 months before eligibility confirmation, or unstable or
    * Uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV)
    * Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Version 5 Grade 2 or higher) or clinically significant ECG abnormalities
    * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >500 msec

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
MRD negativity | Within 12 months after ASCT
  The rate of MRD negativity is determined as the proportion of patients with NGF MRD negativity (10-5 sensitivity level) within 12 months after ASCT using the intention-to-treat principle. For patients who withdraw from the study or are lost to follow up before this timepoint, the best MRD assessment will be considered. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment.

SECONDARY OUTCOMES:
Response rate | 5/6 years
  Response rate (sCR, CR, VGPR, PR, ORR) will be evaluated according to IMWG Response criteria after induction, transplant and maintenance.
TTP (time to progression) | 5/6 years
  TTP will be measured from the date of ICF to the date of first observation of PD, or deaths for PD. Subjects who have not progressed or who withdraw from the study or die from causes other than PD will be censored at the time of the last complete disease assessment. Subjects lost to follow-up will also be censored at the time of last complete disease assessment.
PFS (progression free survival) | 5/6 years
  PFS will be measured from the date of ICF to the date of first observation of PD, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study or who were lost to follow-up will be censored at the time of the last complete disease assessment.
TNT (time to next therapy) | 5/6 years
  TNT will be measured from the date of eligibility confirmation to the date of next anti-myeloma therapy. Death due to any cause before starting therapy will be considered an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. Subjects lost to FU will also be censored at the time of last contact.
PFS2 (progression free survival 2) | 5/6 years
  PFS2 will be measured from the date of ICF to the date of observation of second disease progression (i.e. progression after the second line of therapy) or death to any cause as an event. In case of date of second progression is not available, date of start of third line treatment can be used. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. All subjects who were lost to follow-up prior to the end of the study, have not progressed, and are still alive will also be censored at the time of last contact.
OS (overall survival) | 5/6 years
  OS is defined as the time between ICF date and death, regardless cause of death. Subjects who withdraw consent will be censored at the time of withdrawal. Subjects who are still alive at the cut-off Page 48 of 72 date of final analysis will be censored at the cut-off date. Subjects lost to FU will also be censored at the time of last contact.
DOR (duration of response) | 5/6 years
  DOR is defined as time between first documentation of response (achievement of at least a PR) and PD with deaths owning to causes other than progression not counted, but censored. Responders without disease progression at the cut-off date of final analysis will be censored either at the time of lost to follow-up, at the time of death due to other cause than PD, or at the time of last contact.
Time to PR (time to partial response) | 5/6 years
  Time to PR will be measured from the date of ICF to the date of first observation of PR (Partial Response). Subjects who achieved response better than PR will be consider that PR is achieved. Subjects who withdraw from the study will be censored at the time of the last complete disease assessment. Subjects have not achieved a PR, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to FU will also be censored at the time of last contact.
Time to VGPR (time to very good partial response) | 5/6 years
  Time to VGPR will be measured from the date of ICF to the date of first observation of VGPR (Very Good Partial Response). Subjects who achieved response better than VGPR will be consider that VGPR is achieved. Subjects who withdraw from the study will be censored at the time of the last complete disease assessment. Subjects have not achieved a VGPR, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to FU will also be censored at the time of last contact.
Time to CR (time to complete response) | 5/6 years
  Time to CR will be measured from the date of ICF to the date of first observation of CR (Complete Partial Response). Subjects who achieved response better than CR will be consider that CR is achieved. Subjects who withdraw from the study will be censored at the time of the last complete disease assessment. Subjects have not achieved a CR, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to FU will also be censored at the time of last contact. Difference will be calculated in 30-day months.
Time to sCR (time to stringent complete response) | 5/6 years
  Time to sCR will be measured from the date of ICF to the date of first observation of sCR (stringent Complete Partial Response). Subjects who withdraw from the study will be censored at the time of the last complete disease assessment. Subjects have not achieved a sCR, and are still alive at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to FU will also be censored at the time of last contact. Difference will be calculated in 30-day months.
Rate of 1 year sustained MRD (minimal residue disease) negativity | 5/6 years
  Rate of 1 year sustained MRD negativity by NGF will be also evaluated, and correlated with PFS and OS.
MRD (minimal residue disease) negativity | 5/6 years
  The rate of MRD negativity is determined as the proportion of patients with NGF MRD negativity (10-5 sensitivity level) within 12 months after ASCT using the intention-to-treat principle. For patients who withdraw from the study or are lost to follow up before this timepoint, the best MRD assessment will be considered. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment.
24 months MRD negativity rate | 5/6 years
  The 24 months MRD negativity rate is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level, NGF) after 12 months using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment/sample not adequate.
Analysis of safety | 5/6 years
  The analysis of safety as defined by type, frequency and severity will be done primarily by tabulation of the incidence of Adverse Events as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. In the by-subject analysis, a subject having the same event more than once will be counted only once. Adverse Events will be summarized by worst CTCAE grade.
Dose reduction rate | 5/6 years
  Dose reduction will be done primarily by tabulation of the incidence of dose reduction and causes.
Time to discontinuation of study drug | 5/6 years
  Time to discontinuation will be measured from the date of first dose of study drugs to the date of discontinuation due to AE or Death for AE/SPM. Subjects who discontinued drugs due to PD, or death for cause other than AE/SPM will be considered a competitive event. Subjects has not discontinued, and are still alive and on treatment at the cut-off date of final analysis will be censored at the cut-off date. All subjects who were lost to FU will also be censored at the time of last contact.
Relative dose estimations for each study drugs | 5/6 years
  Relative dose will be evaluated consider the ration between the administered and the planned dose. Relative dose will be estimated for each study drugs.

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (14):
  - AOU Ospedali Riuniti Umberto I, Ancona
  - AOU Policlinico di Bari, Bari
  - AOU di Bologna, Bologna
  - Ospedale di Bolzano - Azienda Sanitaria dell'Alto Adige, Bolzano
  - AOU Policlinico S. Martino, Genova
  - I.R.C.C.S. Ospedale S. Raffaele, Milan
  - AOU Federico II, Napoli
  - AO di Padova, Padua
  - AO di Perugia-Ospedale S. Maria della Misericordia, Perugia
  - Policlinico Umberto I - Università 'Sapienza', Roma
  - AO S. Maria, Terni
  - AOU Città della Salute e della Scienza di Torino, Torino
  - AOU Ospedali Riuniti di Trieste, Trieste
  - Ospedale S. Maria della Misericordia di Udine, Udine